CLINICAL TRIAL: NCT06739564
Title: Dry Needling Vs Ice Packing in Acute Recovery After a Strenuous Effort in Semi-pro Football Players.
Brief Title: Dry Needling and Ice Packing in Recovery.
Acronym: D-NICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, ANTONIO CICCHELLA, Principal Investigator, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tjdxsr029
Record Dates: First submitted 2024-12-03; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Recovery Method; Fatigue Intensity
Keywords: fatigue; recovery; soccer; pain threshold
MeSH Terms: conditions — Fatigue | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dry needling (Experimental): Dry needling on lower limbs
  Interventions: Procedure: DRY NEEDLING
- Ice packing (Experimental): ice packing on lower limbs
  Interventions: Procedure: ICE PACKING
- controls (No Intervention): control group

INTERVENTIONS:
Procedure: ICE PACKING — ICE PACKING ON LOWER LIMB AFTER AN EXHAUSTION EFFORT.
  Arms: Ice packing
Procedure: DRY NEEDLING — DRY NEEDLING ON LOWER LIMB AFTER AN EXHAUSTION TRIAL
  Arms: Dry needling

SUMMARY:
Recovery is a crucial aspect of soccer training. It has been investigated scientifically, but some unclear aspects remain regarding the optimal strategy. Recovery from maximal effort involves both physical and psychological/perceptual aspects (pain, sleep quality), and the definition of recovery is often misleading due to the subjective and objective factors involved. This is a randomized control trial comparing dry needling (DN) to ice packing (ICE) in the acute recovery after an exhaustion running trial in thirty-nine semi-professional soccer players compared to controls. The subjects were assessed before and after the exhaustion tests for sleep, pain perception (Pressure Pain Threshold, PPT), Counter Movement Jump (CMJ), and Surface Muscle Temperature (SMT). We tested 39 semi pro soccer players (males and females).

DETAILED DESCRIPTION:
This is a randomized controlled trial involving thirty-nine subjects: 15 in the control group (CG, 6 females, 9 males), 12 in the ice packing group (ICE, 6 males and 6 females), and 12 in the dry needling group (DN, 6 males and 6 females). Semi-professional players from clubs in Shanghai city participated in the study. Inclusion criteria were not having ongoing or past muscular illness in the last three months and regularly take part in training at least 5 times per week. Exclusion criteria were having an injury in the lower limbs in the last three month and taking any anti-inflammatory or pain killer drugs. The participants gave their informed written consent to participate. The subjects visited the laboratory twice on different days.

After 10 minutes of running at a chosen speed, the subject was tested for VO2max (Cosmed K5, Rome, Italy) on a motorized treadmill (Rodby RL2000, Sweden), starting at a comfortable speed and rising one step of 2 km/h every minute until exhaustion. Once VO2max was assessed, the anaerobic threshold (AT) was determined by the Cosmed software using the V-slope method and was later checked and adjusted by two expert observers . Two days after the VO2max test, the subjects visited the laboratory and performed a trial at AT on the treadmill until exhaustion. The trial was stopped by the subject's signalling exhaustion by raising an arm. Blood lactate was measured twice, after the VO2max test and after 3 minutes from the termination of the exhaustion trial using a lactacidometer (Lactate Pro, Germany) to assess the consistency of effort. Body weight and body fat percentage were measured with a Tanita scale-impedenziometer and body height with a Tanita anthropometer. The groups matched for body height, weight, and body fat percentage.

SMT was measured after the exhaustion trial, and after the recovery procedures. After the exhaustion trial, DN and ICE were performed. Ice packs were applied to the quadriceps, hamstrings, and soleus/gastrocnemius muscles for 20 minutes, and DN was performed by inserting the needles at relevant trigger points of the lower limb. PPT was measured before and after the recovery procedures with an FPX50 pressure gauge (Wagner, USA) on the left and right quadriceps, gastrocnemius medialis, and lateralis. The sequence of the measurements after the exhaustion trial followed the same pre-treatment order. A maximal Counter Movement Jump (CMJ) test (best of 3 trials) was recorded with a video analysis app (My Jump Lab, v.4.2.6).

The choice of latent MTrPs (trigger points) was made according to the following criteria [38]: 1) palpable taut band; 2) hypersensitive spot on the taut band; and 3) palpation with the reproduction of the patient's symptoms that include different sensory sensations, including pain spreading to a distant area, deep pain, dull ache, tingling, or burning pain. If the above three points are satisfied, it is an active trigger point, and if both 1 and 2 were met, but not 3, then it was considered a latent trigger point. The quadriceps (rectus femoris, vastus medialis, and vastus lateralis), tensor fasciae latae, hip adductors (adductor longus, adductor brevis), hip abductors (gluteus medius, gluteus maximus), and gastrocnemius were examined in each subject following a protocol regarding patient and limb positions reproduced from previous studies . Diagnostic criteria were applied by physical therapists with five years of experience with myofascial pain.

After the skin was locally sterilized, the MTrPs were transcutaneously punctured with a 0.30 mm × 40 mm or 0.30 mm × 75 mm sterilized disposable stainless-steel acupuncture needle. During dry needling, the left thumb or two fingers pressed or held the taut band. The right hand was used to quickly insert the needle into the latent MTrPs, then punctured back and forth into the taut band in different directions until a local twitch response was elicited. Once the first local twitch response was obtained, the needle was moved up and down at approximately 1 Hz until no more local twitch responses were elicited. After pulling out the needle, ischemic compression with a finger was applied for 10-30 seconds. The DN insertion was made by a certified Chinese medicine clinician.

To measure SMT, a Manual Infrared Camera (BX20, HK micro, Hangzhou, China) with a sensor resolution of 1024 × 768 pixels was employed, with a measurement range from 0 °C to 250 °C, a display of 230 × 240 pixels, a thermal sensitivity of 80 mK, and an 8-mm lens. The infrared thermography imaging acquisition was performed with the participant standing up in a relaxed position 1 m from the camera. It was measured in a region of interest (ROI) through five infrared thermography images of different muscle sectors for each muscle on the quadriceps and calf muscles on both legs. We considered the max and min temperature and the central value in the ROI (region of interest). After removing the highest and lowest values, the mean of the three measurements was used for data analysis. The SMT can be affected by environment temperature and humidity due to sweating, evaporation and vasoconstriction/vasodilation response. To maintain consistency, we controlled the air temperature and humidity in the lab. Specifically, the room temperature and humidity were kept at 20.0-23.0 °C and 60-75%, respectively . Sleep (light, deep, REM, and total sleep time, in hours) was measured with a sleep monitor (Huawei Band 8) the night before the exhaustion test and after the recovery procedures . RPE (Scale 20 items) and Lactate (Lactate Pro, Germany) were measured two times, after the VO2max and after the exhaustion test at 3 and 5 minutes, and the highest value was retained. RPE and Lactate were used to assess the consistency of the exhaustion trial. The study was conducted according to the guidelines of the Declaration of Helsinki and approved by the Ethics Committee of Tongji University (approval code: tjdxsr029).

ELIGIBILITY:
Inclusion Criteria:

* not having ongoing or past muscular illness in the last three months and regularly take part in training at least 5 times per week.

Exclusion Criteria:

* Exclusion criteria were had an injury in the lower limbs in the last three month and taking any anti-inflammatory or pain killer drugs.

Ages: 19 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-03 (Actual)

PRIMARY OUTCOMES:
Surface muscle temperature in degrees Centigrades. | acute, after a few minutes (20) the data are available. It will be reported in 3 months from the measurement ending.
  SMT was measured after the exhaustion trial, and after the recovery procedures. After the exhaustion trial, DN and ICE were performed. Ice packs were applied to the quadriceps, hamstrings, and soleus/gastrocnemius muscles for 20 minutes, and DN was performed by inserting the needles at relevant trigger points of the lower limb. PPT was measured before and after the recovery procedures with an FPX50 pressure gauge (Wagner, USA) on the left and right quadriceps, gastrocnemius medialis, and lateralis. SMT was measured immediately after ICE and DN in a time frame of 20 minutes from the beginning on test to the end. Final data will be reported in 3 months.
Pressure pain threshold in algometer units scale. | acute, after a few minutes (20) the data are available. It will be reported in 3 months from the measurement ending.
  PPT was measured before and after the recovery procedures with an FPX50 pressure gauge (Wagner, USA) on the left and right quadriceps, gastrocnemius medialis, and lateralis. Time frame: this outcome is evaluated after 20 minutes. Final data will be reported in 3 months. Final data will be reported in 3 months.
Squat Jump in cm | acute, after a few minutes (20) the data are available. It will be reported in 3 months from the measurement ending.
  A maximal Counter Movement Jump (CMJ) test (best of 3 trials) was recorded with a video analysis app (My Jump Lab, v.4.2.6). Time frame: this outcome is evaluated after 30 min from the termination of the test and before the fatigue test. Final data will be reported in 3 months.
Perceived effort in RPE scores | acute, after a few minutes (20) the data are available. It will be reported in 3 months from the measurement ending.
  Borg Rate Perceived Excerption (Scale 20 level: higher the level higher the perceived effort) was measured two times, after the VO2max and after the exhaustion test at 3 and 5 minutes, and the highest value was retained. Evaluated after 1 minutes from the termination of fatigue test. Final data will be reported in 3 months.
Lactate in mm/L (millimoles x liter) | acute, after a few minutes (20) the data are available. It will be reported in 3 months from the measurement ending.
  Lactate (Lactate Pro, Germany) was measured two times, after the VO2max and after the exhaustion test at 3 and 5 minutes, and the highest value was retained. Lactate was used to assess the consistency of the exhaustion trial. Lactate was evaluated at 3 and 5 minutes after the ending of the exhaustion test. Final data will be reported in 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongji University, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: No
PRIVACY

REFERENCES:
- [Background] You S, Shen Y, Liu Q, Cicchella A. Patellofemoral Pain, Q-Angle, and Performance in Female Chinese Collegiate Soccer Players. Medicina (Kaunas). 2023 Mar 16;59(3):589. doi: 10.3390/medicina59030589. PMID 36984590